CLINICAL TRIAL: NCT05212142
Title: A Strategy to Prevent the Recurrence of Dental Disease in Children Receiving Dental Treatment With General Anesthesia: a Randomized Controlled Trial
Brief Title: A Strategy to Prevent the Recurrence of Dental Disease in Children Receiving Dental Treatment With General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HM20023677
Record Dates: First submitted 2022-01-25; First posted 2022-01-27 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Caries
MeSH Terms: interventions — Audiovisual Aids; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional intervention: verbal education (Sham Comparator)
  Interventions: Behavioral: verbal education
- New intervention: verbal education, visual aids, and motivational interviewing (Experimental)
  Interventions: Behavioral: verbal education, visual aids, and motivational interviewing

INTERVENTIONS:
Behavioral: verbal education — Participants will receive oral health anticipatory guidance in the form of verbal and written education alongside the same preventive follow up and recall appointment schedule.
  Arms: Traditional intervention: verbal education
Behavioral: verbal education, visual aids, and motivational interviewing — Participants will receive oral health anticipatory guidance through a combination preventive strategy using motivational interviewing, individualized goal setting, visual aids, and verbal education alongside a preventive follow up and recall appointment schedule
  Arms: New intervention: verbal education, visual aids, and motivational interviewing

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a preventive strategy in increasing return to follow up and recall appointments.

ELIGIBILITY:
Inclusion Criteria:

1. parent with child (patient) planned for dental treatment with general anesthesia (GA)
2. parent of a child (patient) age less than six
3. parent of a child (patient) with health status of healthy (American Society of Anesthesiologists (ASA) I or II).

Exclusion Criteria:

1. parents/guardians who chose not to participate in the study
2. parents who spoke a language other than English or Spanish
3. Parents of a child (patient) with special health care needs or patients of ASA III or IV status

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Change in parental self-efficacy (PSE) | Baseline to 2 weeks
  The PSE questionnaire adapted from an combination of questions developed by Dumka et al. and Johnston & Mash will measure parents perceived self-efficacy in controlling their child's oral health.
Change in parent oral health knowledge | Baseline to 2 weeks
  A questionnaire developed by Alsada et al. will be adapted and used to test parent's knowledge of overall oral health.
Follow up return rate | 2 weeks
  Number of participants who return for follow up in 1 - 2 weeks.
3-month recall return rate | 3 months
  Number of participants who return for follow up in 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jayakumar Jayaraman, DDS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No